CLINICAL TRIAL: NCT04010006
Title: Randomized Controlled Trials Comparing Clinical Outcome of HD Versus 4K Laparoscopy for Gastric Cancer(FUGES-017)
Brief Title: Trials Comparing of HD Versus 4K Laparoscopy for Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Head of gastric surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-017
Record Dates: First submitted 2019-05-09; First posted 2019-07-08 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Laparoscopy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4K Laparoscopic Surgery (Experimental): 4K Laparoscopic Surgery will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: 4K Laparoscopic Surgery
- HD Laparoscopic Surgery (Active Comparator): HD Laparoscopic Surgery will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: HD Laparoscopic Surgery

INTERVENTIONS:
Procedure: 4K Laparoscopic Surgery — 4K Laparoscopic Surgery will be performed for the treatment of patients assigned to this group.
  Arms: 4K Laparoscopic Surgery
Procedure: HD Laparoscopic Surgery — HD Laparoscopic Surgery will be performed for the treatment of patients assigned to this group.
  Arms: HD Laparoscopic Surgery

SUMMARY:
The purpose of this study is to explore the feasibility of 4K Laparoscopic Surgery for Gastric Cancer.

DETAILED DESCRIPTION:
A prospective randomized comparison of HD and 4K laparoscopic surgery for gastric cancer will be performed, to evaluate the clinical value and provide theoretical basis and clinical experience for the extensive application of the 4K laparoscopic technique. The evaluation parameters are perioperative clinical efficacy, postoperative life quality, immune function and 3-year survival and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* (1)Age from over 19 to under 74 years
* (2)cT 1-4a(clinical stage tumor), N0-3, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
* (3)Heart, lungs, kidneys and other vital organs function well, with no obvious surgical contraindications
* (4)Preoperative examination with no distant metastasis, no significantly enlarged lymph nodes around abdominal main artery, and tumor not a direct violation of the pancreas, spleen and other surrounding organs
* (5)American Society of Anesthesiology (ASA) score class I, II, or III
* (6)Written informed consent

Exclusion Criteria:

* (1)Women during pregnancy or breast-feeding
* (2)Severe mental disorder
* (3)History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* (4)Enlarged splenic hilar lymph nodes with integration into a mass and surrounding the blood vessels
* (5)History of unstable angina or myocardial infarction within past six months
* (6)History of cerebrovascular accident within past six months
* (7)History of continuous systematic administration of corticosteroids within one month
* (8)History of previous neoadjuvant chemotherapy or radiotherapy
* (9)T4b tumors
* (10)Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* (11)FEV1(Forced expiratory volume in one second)#50% of predicted values

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
operating time | 1 day
  day

SECONDARY OUTCOMES:
The number of lymph node dissection | 1 day
  number
the number of positive lymph nodes | 1 day
  the number of positive lymph nodes
intraoperative lymph node dissection time | 1 day
  (regional analysis:infrapyloric area lymph node,suprapancreatic area lymph node,splenic hilar area lymph node,cardial area lymph node)
intracavitary anastomosis time | 1 day
  (patients who undergo totally laparoscopic surgery are analyzed)
intraoperative blood loss | 1 day
  ml
intraoperative injury | 1 day
  intraoperative injury
the amount of use of titanium clip | 1 day
  the amount of use of titanium clip
the rate of conversion to laparotomy | 1 day
  the rate of conversion to laparotomy
Time to first ambulation | 10 days
  Time to first ambulation
Time to first flatus | 10 days
  Time to first flatus
Time to first liquid diet | 10 days
  Time to first liquid diet
Time to first soft diet | 10 days
  Time to first soft diet
duration of postoperative hospital stay | 10 days
  duration of postoperative hospital stay
Complication | 30 days;36 months
  (early complications occurred within 30 days after operation): pulmonary infection, incision complication, intestinal obstruction, abdominal infection, anastomotic bleeding, anastomotic fistula, gastric emptying; long term complications (30 days later after operation): anastomotic stenosis, intestinal obstruction, dumping syndrome
The daily highest body temperature before discharge | 7 days
  The daily highest body temperature before discharge
Overall postoperative morbidity and mortality rates | 30 days
  The number of all patients treated with surgery as the denominator and the number of the patients with any intraoperative and postoperative morbidity and mortality as the numerator are used to calculate the proportions.
  Postoperative morbidities are divided into short-term and long-term complications after surgery.
  Short-term is defined as within 30 days of surgery or the first discharge if the hospital stay is > 30 days.
  Long-term is defined as the period from 30 days or more after the operation or the period between first discharge (the hospital days after surgery >30 days) and 3 years after the operation.
  Postoperative mortality: patients whose death was identified according to documented intraoperative observation items, including patients who die within 30 days after surgery (including the 30th day) regardless of the causality between death and surgery, and patients who die more than 30 days after surgery.
Hospitalization expenses | 1 months
  dolloars
3-year disease free survival rate | 36 months
  month
3-year overall survival rate | 36 months
  month

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang Huang, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No